CLINICAL TRIAL: NCT06706518
Title: Systematic Workflow for Pentaspline Pulsed-field Ablation Optimization: Real-world Performance of the 12 COmmandments (12-O) Strategy
Acronym: 12-O strategy
Status: Completed | Type: Observational
Sponsor: Daniel Rodríguez Muñoz (Other)
Responsible Party: Sponsor-Investigator, Daniel Rodríguez Muñoz, Cardiologist, Head of Cardiac Electrophysiology, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: SWEET-Shot
Record Dates: First submitted 2024-11-25; First posted 2024-11-26 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (Paroxysmal); Atrial Fibrillation (AF); Ablation of Atrial Fibrillation
Keywords: Pulmonary Vein ablation; Atrial Fibrillation; SWEET Strategy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Paroxysmal or persistent AF diagnosis and a PVI clinical indication: Patients >18 years old, with a diagnosis of paroxysmal or persistent AF and a clinical indication to undergo PVI
  Interventions: Procedure: Single-shot ablation technologies

INTERVENTIONS:
Procedure: Single-shot ablation technologies — Comparison of fluoroscopy time and dose-area product (DAP) between different single-shot ablation technologies.
  * PolarFit balloon catheter with adjustable diameter 28 to 31 mm. This catheter will be used in patients with persistent AF and dilated left atrium, where the ability to encompass more of the atrial myocardium at the level of the antrum of the pulmonary veins allows a greater number of potential AF perpetuating regions to be covered.
  * ArcticFront Advance Pro 28 mm diameter balloon catheter*.
  * 28 mm diameter PolarX balloon catheter*.

SUMMARY:
In our center we have developed a systematic approach to pulmonary vein cryoablation (SWEET Cryo strategy) that has been shown to reduce radiation during the procedure substantially without increasing the cost associated with the procedure. This study, however, has been done on the basis of pulmonary vein cryoablation technology available on the market in the last 10 years. The appearance of new cryoablation technologies (greater degree of sheath deflection, greater balloon catheter complexity, balloon with expandable diameter) and new energy sources, such as pulsed electric field ablation or "electroporation" for "single shot" ablation, which significantly modify the workflow during the procedure, raises the question of whether the strategy developed and validated in our center is applicable to these other technologies, which are already being used in our center.

Specifically in relation to pulsed electric field ablation, the question arises as to the impact that a fluoroscopy reduction strategy may have on clinical outcomes. This is due to the need for catheter contact with the tissue, which in the case of cryoablation is guaranteed by verification of vein occlusion (contrast retention) but which in this new technology is not, since the vein is not occluded and therefore there is no possibility of verification of contact with the tissue by this means. Thus, the use of X-rays is the best way to estimate the degree of contact, which determines the durability of the treatment in the long term. In this regard, there are discordant data in different series of the initial application of this technology. While the initial evidence showed between 96 and 100% durability of pulmonary vein isolation, recent registries on the real-life application of this technology show reconnection of at least one pulmonary vein in 28% of patients undergoing re-intervention for clinical recurrence of atrial fibrillation.

DETAILED DESCRIPTION:
The primary objective of this study is the comparison of fluoroscopy time and dose-area product (DAP) between the different single-shot ablation technologies available in our center after application of the "SWEET" strategy for reducing X-ray exposure. Secondary objectives are efficacy and safety outcomes.

The hypothesis is that this systematic approach allows a significant reduction in the radiation used in this procedure in all single-shot techniques, while maintaining its efficacy and safety.

The secondary hypothesis is that the reduction of fluoroscopy during the procedure does not obtain worse results in terms of durability of pulmonary vein isolation with respect to what is reported in routine clinical practice registries.

Taking into account previous data from the experience in our center, it is considered that, in order to obtain a representative sample, not conditioned by extreme values of cases with punctual particularities, of fluoroscopy and PDA time values, data from 40 patients with each technique should be collected and analyzed:

* 31 mm Farawave catheter ablation using pulsed electric fields. This catheter will be used in patients with resting heart rate >70 bpm in whom it is estimated that there is less likely to be a vagotonic component in AF perpetuating mechanisms, since the energy source does not act on cardiac ganglionic plexuses.
* PolarFit balloon catheter with adjustable diameter 28 to 31 mm. This catheter will be used in patients with persistent AF and dilated left atrium, where the ability to encompass more of the atrial myocardium at the level of the antrum of the pulmonary veins allows a greater number of potential AF perpetuating regions to be covered.
* ArcticFront Advance Pro 28 mm diameter balloon catheter*.
* 28 mm diameter PolarX balloon catheter*.

  * These last two catheters will be used indistinctly in patients who do not present the previously mentioned characteristics-.

Ablation will be performed according to standard clinical practice, with the only difference being the application of this protocol to minimize the use of radiation.

Patient demographic variables will be collected, preserving the anonymity of the data by assigning a specific code for the study and not linked to the patient's medical history number or other identifying data.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old, with a diagnosis of paroxysmal or persistent AF and a clinical indication to undergo PVI were included

Exclusion Criteria:

* prior PVI or left atrial linear ablation
* severe frailty or life expectancy <1 year
* unwillingness or inability to provide informed consent
* ablation at sites beyond PVI
* contraindication or intolerance to heparin
* presence of left atrial thrombus
* congenital heart disease
* pregnancy, ongoing or planned in the following 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing PVI with a diagnosis of paroxysmal or persistent AF recruited in single tertiary university hospital: Hospital 12 de Octubre
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy time during ablation procedure (min) | It is assessed through procedure time, measured in minutes
  Co-primary efficacy endpoint
Durable PVI effect | After 90 days of first PVI ablation
  Co-primary efficacy endpoint. In the subgroup of patients undergoing pulsed electric field ablation (31 mm Farawave catheter), a second procedure for re-mapping of the pulmonary veins will be performed no earlier than 90 days after the initial procedure. This procedure will check if the pulmonary veins remain isolated.
Cardiac Major Adverse Events | In the first 30 days following either the index or remapping procedures
  Primary safety endpoint is a composite of major adverse events (AEs) including cardiac perforation, tamponade, stroke or transient ischemic attack, peripheral thromboembolic event, vascular complications requiring intervention, myocardial infarction or death occurring in the first 30 days following either the index or remapping procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain